CLINICAL TRIAL: NCT02563600
Title: Effect of Brief-tele Support on Attendance at Physiotherapy Sessions for Pelvic Floor Dysfunctions
Brief Title: Effect of Brief-tele Support on Attendance at Physiotherapy Sessions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Abertawe Bro Morgannwg University Health Board (Other)
Responsible Party: Principal Investigator, Prof Phil Reed, Professor Phil Reed, Swansea University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: SwanseaU
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Floor Dysfunctions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-letter telephone call (Experimental): A brief 10 min telephone call to patients on waiting list prior to receipt of appointment invitation letter.
  Interventions: Behavioral: Pre-letter telephone call.
- Post-letter telephone call (Experimental): A brief 10 min telephone call to patients on waiting list prior to receipt of appointment invitation letter.
  Interventions: Behavioral: Post-letter telephone call
- No telephone call (No Intervention): No telephone call made to patient.

INTERVENTIONS:
Behavioral: Pre-letter telephone call. — A brief 2-10 min telephone call made to the patient prior to receipt of appointment invitation letter.
  Arms: Pre-letter telephone call
Behavioral: Post-letter telephone call — A brief 2-10 min telephone call made to the patient after receipt of appointment invitation letter.
  Arms: Post-letter telephone call

SUMMARY:
Patients on the waiting list for physiotherapy treatment for pelvic floor dysfunction will be randomly divided into three groups:

* a group that gets a telephone call before their invitation letter is sent.
* a group that gets a telephone call after their invitation letter is sent.
* a group that does not receive a telephone call.

The phone call is a brief 5-10 minute call, which will be semi-structured. It will remind the patient of their appointment time, it will outline what the treatment involves and highlight the potential benefits and drawbacks, and allow the patient to ask questions about the treatment.

DETAILED DESCRIPTION:
Aims:

The research aims to assess the impact of a brief telephone call to patients with pelvic floor problems who are on a waiting list for physiotherapy treatment. Non-attendance at sessions currently runs at about 50%, and steps to reduce this would be beneficial to patient health and NHS efficiency.

Participants and Recruitment:

Consecutive patients who have been referred for physiotherapy treatment for pelvic floor dysfunction will be asked if they would like to participate in the study. The initial approach will be made through a letter, which will give information about the study, and will make clear that their treatment will not depend on their participation in the study.

Patients on the waiting list for physiotherapy treatment for pelvic floor dysfunction will be randomly divided into three groups:

* a group that gets a telephone call before their invitation letter is sent
* a group that gets a telephone call after their invitation letter is sent
* a group that does not receive a telephone call.

The phone call is a brief 5-10 minute call, which will be semi-structured. It will remind the patient of their appointment time, it will outline what the treatment involves and highlight the potential benefits and drawbacks, and allow the patient to ask questions about the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women on waiting list for pelvic floor dysfunction
* over 18 years old

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who attended their first schedules physiotherapy session | At first scheduled physiotherapy session which will be two to four weeks following the invitation letter

CONTACTS AND LOCATIONS:
Overall Officials: Phil Reed, D.Phil., Principal Investigator — Swansea University
Locations (1):
- Singleton Hospital, Swansea, United Kingdom

REFERENCES:
- [Derived] Osborne LA, Whittall CM, Emanuel R, Emery S, Reed P. Randomized Controlled Trial of the Effect of a Brief Telephone Support Intervention on Initial Attendance at Physiotherapy Group Sessions for Pelvic Floor Problems. Arch Phys Med Rehabil. 2017 Nov;98(11):2247-2252. doi: 10.1016/j.apmr.2017.03.033. Epub 2017 May 17. PMID 28526481